CLINICAL TRIAL: NCT05791864
Title: A First-in-Human, Open-Label, Dose-Escalation Study to Evaluate the Safety and Tolerability of Gene Therapy With TTX-381 for the Ocular Manifestations Associated With Neuronal Ceroid Lipofuscinosis Type 2 (CLN2) Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tern Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TTX-381-1102; 2021-000173-92 (EudraCT Number)
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-02

CONDITIONS: Neuronal Ceroid Lipofuscinosis Type 2
Keywords: CLN2; Batten Disease; Gene Therapy
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — Genetic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In order to minimize the effect of potential bias, wherever possible, endpoints will be measured or interpreted by masked evaluators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Main Treatment Arm (Experimental): 2×10^10 GC/eye
  Interventions: Genetic: TTX-381
- Cohort 2: Main Treatment Arm (Experimental): 6×10^10 GC/eye
  Interventions: Genetic: TTX-381
- Expansion Cohort (Experimental): Expansion cohort, dose level 2×10^10 GC/eye as determined by Independent Data Monitoring Committee.
  Interventions: Genetic: TTX-381

INTERVENTIONS:
Genetic: TTX-381 — One time subretinal dose in study eye
  Other Names: Gene Therapy (AAV9.CB7.hCLN2)

SUMMARY:
This is a first-in-human, open-label, single ascending dose study of TTX-381 for the treatment of ocular manifestations of CLN2 (Batten disease).

DETAILED DESCRIPTION:
This is a first-in-human, open-label, single ascending dose study of TTX-381, a gene therapy for the potential treatment of ocular manifestations of CLN2 (Batten disease). TTX-381 is being studied as a potential treatment of ocular manifestations of neuronal ceroid lipofuscinosis type 2 (CLN2) disease. Children with CLN2 disease have a non-working gene (set of instructions) that causes an enzyme called tripeptidyl-peptidase 1 (TPP1) to be missing or not working in their bodies. Without enough TPP1, cells cannot break down certain molecules in the body, so these storage materials build up and start to hurt the body, particularly the central nervous system (the brain and spine) and retinal cells (eyes); cause seizures; and change how children with CLN2 disease grow, act, think, and see. After eligibility has been confirmed, the participant's eyes will be assigned as the treated eye and the control fellow eye. Due to the symmetry in the clinical course of CLN2 ocular disease, untreated fellow eyes will serve as controls for the contralateral, treated eyes. Participants will be followed in this study for 5 years after TTX-381 administration.

ELIGIBILITY:
Inclusion Criteria:

A participant is eligible to be included in the study only if all of the following criteria apply:

* Has biallelic CLN2 mutations.
* Has decreased leukocyte TPP1 activity.
* Has clinical signs or symptoms consistent with CLN2 disease (eg, developmental delay, developmental decline, seizure, vision loss, or other signs/symptoms) OR an older sibling with confirmed CLN2 diagnosis.
* Is currently receiving biweekly ICV ERT treatment with cerliponase alfa.
* Meets the following baseline disease condition according to age and CRT as assessed by SD-OCT and confirmed by CRC:

Participants in the phase of accelerated decline in CRT:

1. CRT at baseline ≤210 μm and
2. CRT at baseline ≥140 μm in both eyes and
3. Age ≤84 months,

   * Is willing to adhere to the protocol and 5-year visit schedule.
   * Sexually active female participants of childbearing potential (following menarche) or fertile male participants (following puberty) must be willing to use a medically accepted form of contraception from Screening Visit 2 until 6 weeks after vector administration.

OR

* Was previously administered TTX-381.
* Upon retrospective review, met the above criteria at the time of administration of TTX-381. IDMC may consider exceptions to this when weighing whether to retrospectively enroll a participant who has received TTX-381.
* Has been recommended for enrollment into the clinical trial by IDMC

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any ocular or systemic condition that, in the opinion of the investigator, would prevent administration and evaluation of the investigational product or interpretation of participant safety or study results (eg, significant lens or corneal opacities, glaucoma, amblyopia, gross retinal anatomical abnormality, etc).
* Difference in screening CRT measurement between the right and left eye >10μm.
* Prior Grade 3 or 4 hypersensitivity reaction, eg, bronchospasm and hypotension requiring intravenous treatment, cardiac dysfunction, anaphylaxis to ICV cerliponase alfa infusion.
* Any other contraindication to the administration of ICV cerliponase alfa, including ventriculo-peritoneal shunt, acute intracerebroventricular access device leakage, device failure, or device-related infection that would impact ability to receive ICV cerliponase alfa.
* Prior participation in a gene therapy study. A subject who has received subretinal TTX-381 under a compassionate use protocol may be enrolled if the PI, Medical Monitor, and Sponsor all agree that he/she can safely and successfully participate in the study and the IDMC has approved their enrollment.
* Prior participation in another ocular clinical trial, except an intravitreal cerliponase alfa trial where a subject has received a maximum of 3 injections and the PI, Medical Monitor, and Sponsor all agree that he/she can safely and successfully participate in the study after a washout period of 3 or more months.
* Prior intraocular injections of any kind, with the following two exceptions. A subject who has received a maximum of 3 intravitreal injections of cerliponase alfa may be enrolled in the study if the PI, Medical Monitor, and Sponsor all agree that he/she can safely and successfully participate in the study after a washout period of 3 or more months. A subject who has received subretinal TTX-381 under a compassionate use protocol may be enrolled if the PI, Medical Monitor, and Sponsor all agree that he/she can safely and successfully participate in the study and the IDMC has approved their enrollment.
* Participation in a nonocular clinical study with an investigational drug in the past 6 months prior to screening, except for intracerebroventricular cerliponase alfa.
* Ocular surgery within the prior 6 months except as above for subretinal TTX-381 administration.
* Prior bone marrow transplant. Use of the following medications within the 30 days prior to treatment: gemfibrozil, mycophenolate, prednisone or other steroids for the intended purpose of treating NCL (not including asthma indications), flupirtine.
* Known sensitivity or contraindications to medications planned for use in the peri-operative period.
* Contraindications to systemic immunosuppression.
* Severe renal insufficiency as determined by an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, based on creatinine, at Screening. If the laboratory determines that the creatinine level is less than the lower limit of assay validation or detection, then the lowest limit cutoff value will be used to estimate eGFR.
* Severe hepatic insufficiency as determined by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN) or total bilirubin > 1.5 × ULN at Screening Visit 1, unless the subject has a previously known history of Gilbert's syndrome and a fractionated bilirubin that shows conjugated bilirubin < 35% of total bilirubin.
* Mutations in another CLN gene.
* Mutation in another gene associated with inherited retinal disease.
* Contraindications to intraocular surgery (eg, severe coagulopathy).
* Positive urine pregnancy test at Screening (applying only to females of childbearing potential).
* Any other condition that would not allow the potential participant to complete follow-up examinations during the study or, in the opinion of the investigator, makes the potential participant unsuitable for the study.
* The participant had a positive polymerase chain reaction (PCR) viral test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV2 PCR) within the last 4 weeks before signing the informed consent form (ICF) or has persistent coronavirus disease (COVID-19) symptoms regardless of when the last SARS-CoV2 PCR viral test was performed or when the infection occurred.

Ages: 12 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Ocular and overall AE and SAEs through Day 360 | 360 days
  To evaluate the safety and tolerability of TTX-381 through Day 360 in participants with Neuronal Ceroid Lipofuscinosis Type 2 (CLN2) disease

SECONDARY OUTCOMES:
To evaluate the effect of TTX-381 on area of EZ loss | Day 180, Day 360
  To evaluate the effect of TTX-381 on area of EZ loss as measured by SD-OCT
To evaluate the effect of TTX-381 on central subfield photoreceptor layer thickness | Day 180, Day 360
  To evaluate the effect of TTX-381 on central subfield photoreceptor layer thickness as measured by SD-OCT
To measure TTX-381 transgene product (tripeptidyl peptidase 1 [TPP1]) in aqueous humor | Day 90, Day 360
  To measure TTX-381 transgene product (tripeptidyl peptidase 1 [TPP1]) in aqueous humor
To evaluate shedding of TTX-381 in urine and tears | Day 360
  To evaluate shedding of TTX-381 in urine and tears

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Hamburg-Eppendorf (UKE)- Childrens Hospital, Hamburg, Germany
- Greater Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No